CLINICAL TRIAL: NCT07098624
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Arm, Single-Centre, Clinical Study to Evaluate the Safety and Efficacy of Intake of ACV Moringa on the Degree of Weight Change in Overweight and Class I Obese Study Participants.
Brief Title: Clinical Study to Assess the Safety and Efficacy of ACV Moringa Effervescent Tablet Intake on Weight Management in Overweight and Class I Obese Study Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Zywie Ventures Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB250004-ZV
Record Dates: First submitted 2025-07-17; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Obese or Overweight Healthy Volunteers
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACV Moringa Effervescent Tablets 4.3 g (Experimental): Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Twice daily, once before lunch and once before dinner Storage condition: Room temperature (15°C to 30°C) Route of Administration: Oral
  Interventions: Other: Placebo Effervescent Tablets 4.3 g
- Placebo Effervescent Tablets 4.3 g (Placebo Comparator): Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Twice daily, once before lunch and once before dinner Storage condition: Room temperature (15°C to 30°C) Route of Administration: Oral
  Interventions: Other: ACV Moringa Effervescent Tablets 4.3 g

INTERVENTIONS:
Other: ACV Moringa Effervescent Tablets 4.3 g — Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Twice daily, once before lunch and once before dinner Storage condition: Room temperature (15°C to 30°C) Route of Administration: Oral
  Arms: Placebo Effervescent Tablets 4.3 g
Other: Placebo Effervescent Tablets 4.3 g — Mode of Usage: Dissolve one effervescent tablet in a full glass of water in 200 mL. Allow it to fully dissolve before consuming. For best results, consume the solution immediately after preparation before the fizz ends.
  Frequency: Twice daily, once before lunch and once before dinner Storage condition: Room temperature (15°C to 30°C) Route of Administration: Oral
  Arms: ACV Moringa Effervescent Tablets 4.3 g

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Two-Arm, Single-Centre, Clinical Study to Evaluate the Safety and Efficacy of Intake of ACV Moringa on the Degree of Weight Change in Overweight and Class I Obese Study Participants

DETAILED DESCRIPTION:
This is randomized, double-blinded, single-centre placebo-controlled, two-arms, clinical safety and efficacy study on Overweight and Obese (Class-I) subjects to evaluate the degree of weight change by regular intake of ACV Moringa.

A total of 66 participants (33 Subjects per Test Treatment), including males and non-pregnant, non-lactating females aged between 18 and 65 years, who are overweight/ obese class-I subjects will be enrolled in the study. Participants will be randomized in a 1:1 ratio to receive either Treatment A or Treatment B. The study aims to complete evaluation for 46 participants (23 Subjects per Test Treatment) for the study.

The potential subjects will be screened on the basis of the inclusion and exclusion criteria only after obtaining the written informed consent from the subjects. Subjects will be pre-screened by the Screening Department at NovoBliss Research based on their Body Mass Index (BMI). Subjects will be called contacted telephonically by the recruiting department prior to the enrolment visit. The subject will be requested to bring any previous medications and relevant laboratory reports on the day of the study visit. The subject will be asked to bring the past medications or laboratory reports along with on the study visit day.

The subjects will be instructed to visit the facility as per the below visits:

* Pre-screening
* Visit 01 (Within 30 Days from Day 01): Screening, ICD Obtained, Screening Lab
* Visit 02 (Day 01): Enrolment, Baseline Evaluations, Randomization, Test Treatment phase
* Visit 03 (Day 45 +2 Days): Evaluations, Test Treatment phase
* Visit 04 (Day 90 +2 Days): Final Evaluations, End of Study
* Telephonic Follow-up: A structured telephonic follow-up schedule as mentioned below will be implemented to ensure adherence to study instruction, including diet restrictions and exercise routines. Additionally, daily text messages reminders will be sent to all enrolled subjects.

  * Daily diet adherence reminders will be sent at 8:00 AM (± 2 hours).
  * Daily exercise adherence reminders will also be sent at 8:00 AM (± 2 hours).
  * Weekly digital check-ins will be conducted via the mobile app every Friday. Assessments of efficacy parameters before the administration of the Test Treatments will be done one Day 01 and after the Test Treatment administration will be done on Day 45 (+2 Days) and 90 (+ 2 Days).

Parameters include Anthropometric Parameters, Body composition, Athletic Endurance, Glycemic Parameters, Lipid Metabolism, Metabolic Markers, Inflammatory Biomarkers, Craving Control Biomarkers, Subjective Evaluation, Hematological Profile, Serum Biochemistry

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18- 65 years (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Females of childbearing potential must have a self-reported negative urine pregnancy.
4. Female of childbearing potential must have a reported negative pregnancy during screening and the end of the study
5. Subject is in good general health as determined by the Investigator on the basis of medical history.
6. Subjects who are classified as overweight (BMI 25.0-29.9 kg/m²) or as having Class I obesity (BMI 30.0-34.9 kg/m²).
7. Subjects with a total body fat percentage exceeding 25% for men and 30% for women using Bioimpedance test.
8. Subject is willing to forgo liposuction procedures or any weight loss therapy 3 months prior to and for the duration of the study.
9. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
10. If the female subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
11. If currently using hormonal contraception, has been using this form of contraception for at least 6 months and agrees to continue using the same contraception for the duration of the study.
12. Subject who agree to consume a vegetarian/non-vegetarian diet of approximately 2000 kcal/day (14% protein, 25%Fat and 61% carbohydrate).
13. Subjects willing to follow the given diet and maintain their physical activity by a Diet and physical activity diary.
14. Subjects must possess an Android smartphone to facilitate daily app login and study-related activities.
15. Subjects are willing to give written informed consent and are willing to follow the study procedure.
16. Subjects who commit not to use any other medication for weight management other than the test treatment for the entire duration of the study.
17. Willing to use test treatment throughout the study period.
18. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.

Exclusion Criteria:

1. Subjects BMI is between less than 25 and greater than 35 kg/m2.
2. Subjects having past or present history or clinically significant findings indicating cardiovascular disease, type 2 diabetes mellitus, hypertension, endocrine, pulmonary, neurological or psychological disorders, hypo or hyperthyroidism and renal disorders.
3. Subjects with a history of gastrointestinal disorders, including chronic gastritis, gastric discomfort, or any diagnosed gastrointestinal conditions.
4. Subjects having drug and alcohol abuse.
5. Smokers and tobacco users.
6. Subjects having more than 5 kg variation in body weight within 3 months before study entry.
7. Subjects using other weight loss medications, as well as stimulants, laxatives or diuretics taken solely for the purpose of weight loss.
8. Undergone surgery before 30 days of screening or planning to undergo surgery within the study period.
9. Subjects having chronic diarrhoeal disorders, cancer, hepatic dysfunction, and human immunodeficiency virus (HIV) infection.
10. Participation in other drugs, investigational medicinal product, any herbal products and/or cosmetics intended to weight loss clinical trials within 3 months before enrolment in this trial.
11. Any other diseases/co-morbidity that is considered by the Investigator as an exclusion.
12. With severe hepatic and/or renal impairment, liver enzyme level (ALT and/or AST) is greater than 2.5 times the upper normal limit.
13. Taking antibiotic therapy, anti-depressant treatment or treatment related to anxiety in the month preceding the study,
14. Taking anti-depressant treatment or treatment related to anxiety Subject in a state of depression.
15. Non-stable weight during the last 6 months (>5% change in total weight)
16. Consuming food supplements or functional foods known to have an influence on weight management in the month preceding the inclusion and/or likely to take during the test
17. Following or having followed a hypocaloric diet (energy intake <1,500 kCal/day) in the month preceding inclusion and/or likely to undertake this diet during the test.
18. Diagnosed eating disorders (bulimia, anorexia nervosa, vomiting),
19. Using topical anti-cellulite treatments.
20. Pregnant or breastfeeding or planning to become pregnant during the study period.
21. Subject has a history of chronic illness which may influence the cutaneous state.
22. Subjects participating in other similar nutraceuticals, food, supplemental or therapeutic trials within the last four weeks.
23. Any other condition which could warrant exclusion from the study, as per the Investigator's discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-10-24 (Estimated); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
Change in body weight using calibrated weighing machine | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in body weight in Kg assessed within each treatment group and across treatment groups

SECONDARY OUTCOMES:
Change in Anthropometric Parameters using calibrated measuring tape | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in Anthropometric Parameters (Body weight in kg Waist circumference in cm Hip circumference in cm Height in meter and BMI) assessed within each treatment group and across treatment groups.
Change in total Fat percentage using Bioimpedance Test | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in total Fat percentage assessed within each treatment group and across treatment groups
Change in VO2 Max using Treadmill Walking Test | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in VO2 Max (mL/kg/min) assessed within each treatment group and across treatment groups.
Change in Apolipoprotein - ApoA, ApoB | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in Apolipoprotein (mg/dL) - ApoA, ApoB assessed within each treatment group and across treatment groups.
Change in carbohydrate metabolism through Serum Blood Glucose and PPBG | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in carbohydrate metabolism (mg/dL or mmol/L) assessed within each treatment group and across treatment groups.
Change in Lipid metabolism through Total Cholesterol, HDL, LDL, Triglycerides | visit 01 (30 Days from Day 01) Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in Lipid metabolism (mg/dL or mmol/L) assessed within each treatment group and across treatment groups.
Change in Fatty Acid Oxidation Rate through Beta-hydroxybutyrate | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in Fatty Acid Oxidation Rate (mmol/L) assessed within each treatment group and across treatment groups.
Change in Metabolic Biomarkers through HOMA-IR | Day 01 (pre-treatment), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in Metabolic Biomarkers assessed within each treatment group and across treatment groups.
Change in Inflammatory Biomarkers through IL-6, CRP | Day 01 (pre-treatment), Day 45 (+2 days), and Day 90 (+2 days)
  To assess the efficacy of test treatment by evaluating change in Inflammatory Biomarkers (IL-6 -pg/mL and CRP- mg/L) assessed within each treatment group and across treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, Principal Investigator — NovoBliss Research Pvt Ltd

IPD SHARING:
Plan to Share IPD: No